CLINICAL TRIAL: NCT00641238
Title: Clinical Follow-up of Patients Treated With Radiofrequency Ablation of Lung Masses.
Brief Title: Outcome of Patients With Lung Masses Who Are Treated With Radiofrequency Ablation (RFA)
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Ernest Scalzetti, MD, State University of New York - Upstate Medical University
Other Study IDs: SUNYUMU 4886
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Early stage NSCLC: Early stage non-small cell lung cancer
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Radiofrequency ablation — Radiofrequency ablation

SUMMARY:
We are collecting clinical notes and results of imaging studies (CT and PET scans) from referring physicians who follow the clinical status of patients treated with radiofrequency ablation (RFA). The research objective is to determine whether the patients with (RFA) remain alive, and whether they are in remission or have progressive/ recurrent malignancy

DETAILED DESCRIPTION:
Radiofrequency ablation (RFA) is a relatively new treatment for localized forms of cancer. It requires that a device called a needle-electrode be placed in the tumor. Radiofrequency energy can be passed through this needle-electrode that heats the tissue surrounding the needle tip. If the heating effect is intense enough and maintained for a long enough period of time, the cells in the treated area will be destroyed. RFA has been used in the lung to treat metastases from cancers originating in other sites, and cancers other than small cell carcinoma (Non-small cell lung cancer, NSCLC) that arise in the lung itself.

Pre-treatment assessment includes evaluation of the patient and the tumor itself; this determines whether the patient meets the entry criteria. These criteria are:

* Patient has a biopsy-proven NSCLC, with no other sites of disease, and with a tumor small enough to treat (usually <4 cm). Clinical stage I NSCLC.
* Patient is not a candidate for surgical removal of the cancer, or refused surgery.
* Patient is not a candidate for radiation therapy, or refused radiation therapy.
* Patient has > 6 month life expectancy. The procedure is performed similar to a needle biopsy of the lung, under CT guidance. Placement of the needle-electrode is similar to needle placement for CT-guided biopsy. Appropriate positioning of the needle-electrode is confirmed by CT imaging. Radiofrequency energy is applied to the needle-electrode and the tissue is monitored continuously for electrical changes that indicate tissue destruction. After completion of the treatment, the needle-electrode is removed. The patient is followed for at least three hours prior to discharge. Complications that can be discovered at this time are pulmonary hemorrhage (bleeding in the lung) and pneumothorax (leakage of air from the lung at the site of needle puncture). Subsequent follow-up usually consists of a CT scan at three months and six months after the RFA, and then at six month intervals after that, to see whether the tumor successfully has been transformed into a scar, or continues to grow.

This follow-up is conducted by the referring physician, who may not be associated with this institution. We gather and record this follow-up information until the patient dies, has documented recurrence of the cancer, or completes five years of post- treatment observation. In the cases of recurrence, we also determine whether the tumor is re-growing at the treatment site, or at distant sites that appeared to be uninvolved at the time of treatment.

Statistical analysis will be performed using de-identified patient data. Measures of interest include lifetable determination of median survival and 5-year overall survival. Patients will undergo no study-related procedures during the follow-up period. Chemotherapy given at any time following RFA, at the discretion of a medical oncologist, will not result in exclusion of the patient from analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung masses
* Patients who consent to radiofrequency ablation of mass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical stage I NSCLC that are treated with Radiofrequency ablation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2004-03 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 5 years after diagnosis of NSCLC

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Scalzetti, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- Upstate Medical University, Syracuse, New York, United States